CLINICAL TRIAL: NCT05073640
Title: Pentoxifylline Add-on Therapy for Schizophrenia: A Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Pentoxifylline Add-on Therapy for Schizophrenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mazra Mental Health Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-019-MZR
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline (Active Comparator): Pentoxifylline (Oxopurin 400 mg)
  Interventions: Drug: Oxopurin
- Placebo (Placebo Comparator): Placebo (105 mg Lactose and 510 mg Dextrose)
  Interventions: Drug: Oxopurin

INTERVENTIONS:
Drug: Oxopurin — Subjects will receive two capsules per day.
  Other Names: Pentoxifylline

SUMMARY:
The etiology and pathogenesis of schizophrenia remain unclear. The immune dysfunction hypothesis for schizophrenia has attracted increasing attention from researchers, and substantial evidence suggested that the levels of TNF-α and other cytokines are markedly elevated in patients with schizophrenia. The investigators aim to evaluate the adjuvant therapeutic effect of Pentoxifylline, a TNF-α inhibitor that crosses the blood-brain barrier, in a randomized, double-blind, 6-week trial. Individuals with schizophrenia will receive either Pentoxifylline or a matching placebo as an add-on treatment to antipsychotic agents. Subjects' positive and negative symptoms and plasma concentration of neuroinflammatory markers will be monitored at baseline and every two weeks until the end of the trial.

DETAILED DESCRIPTION:
Ninety schizophrenic patients will be randomized to a Pentoxifylline (400 mg twice a day) or placebo treatment for six weeks. Pentoxifylline and placebo will be added to the current antipsychotic drug treatment. Participants will be asked to fill a socio-demographic questionnaire and to undergo a clinical differential diagnosis using the Symptoms Check List (SCL)-90, Clinical Global Impression (CGI), positive and negative symptoms scale (PANSS), and Hamilton depression rating scale (HAM-D). Following baseline evaluation, participants will be monitored for symptoms every two weeks until the end of the trial (overall three visits) using CGI, PANSS, and HAM-D. Adverse effects will be documented every visit using the Treatment Emergent Symptom Scale. Finally, yet importantly, a blood sample will be collected at baseline and every two weeks until the end of the trial to study the treatment effect on inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the DSM-V criteria for schizophrenia spectrum disorders.
2. Clinical Global Impression (CGI) score ≥ 4 and ≤ 6 at screening.
3. Initiated treatment with a stable dosage of typical and/or atypical antipsychotic medication for at least four weeks.

Exclusion Criteria:

1. Previous sensitivity to pentoxifylline (PTF).
2. Chronic immune and/or inflammatory diseases (such as rheumatoid arthritis, systemic lupus erythematosus, chronic inflammatory bowel disease).
3. Consumption for > 3 consecutive days of any immune-modulating or anti-inflammatory drug in the last month.
4. Current active and persistent substance and/or alcohol abuse.
5. Any severe, unstable medical condition (e.g., cardiovascular disorders, diabetes mellitus, respiratory diseases, cancer).
6. Obesity (body mass index > 30).
7. Cognitive dysfunction such as retardation.
8. Known or suspected pregnancy or breastfeeding women.
9. Lactose intolerance or sensitivity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-20 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Positive and negative symptoms | Subjects will be monitored at baseline and every two weeks for six weeks
  Improvement in positive and negative symptoms (Changes in PANSS rates)

SECONDARY OUTCOMES:
Depressive symptoms | Subjects will be monitored at baseline and every two weeks for six weeks
  Changes in HAM-D rates

CONTACTS AND LOCATIONS:
Locations (1):
- Mazor MHC, Acre, Israel

IPD SHARING:
Plan to Share IPD: Undecided